CLINICAL TRIAL: NCT03784274
Title: Exploration of Pneumonia Related Policy Formation and Implementation in Pakistan
Brief Title: Pneumonia Policy Formation in Pakistan
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Maternal, Neonatal and Child Health Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: AC18007
Record Dates: First submitted 2018-11-26; First posted 2018-12-21 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Pneumonia; Childhood Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stakeholders: Key stakeholders involved program and policy making
  Interventions: Behavioral: Stakeholder analysis

INTERVENTIONS:
Behavioral: Stakeholder analysis — • INCLUSION CRITERIA FOR NET MAPPING ACTIVITIES: Those respondents who are directly involved or knowledgeable about pneumonia related policy environment in the country/province.
  * Respondents who consent to participate in the study.
  * Respondents belonging to Sindh, Punjab, Baluchistan, KPK and Islamabad.
  EXCLUSION CRITERIA:
  • Respondents belonging to Gilgit-Baltistan (GB), Azad Jammu and Kashmir (AJK) and Federally Administered Tribal Area (FATA). Reasons of their exclusion are newly developed governance system (GB), separate governance (AJK) and security threat (FATA).

SUMMARY:
In Pakistan, numerous policies have been formulated in the past on pneumonia management translated into various programs. However, despite completion, the state of pneumonia mortality remains unchanged as no sustainable solutions have been yielded by these programs. This is probably because there was no ownership of these policies and programs at the provincial, district and community level. We, therefore, plan to understand pneumonia related policy environment within Pakistan to identify gaps in this system through a two phased study. The first will be qualitative with key informant interviews conducted from relevant stakeholders, e.g, policy makers, practitioners, academicians, researchers etc., to understand how policies are conceptualized. Data will be analyzed through an integrated approach in a software. The second phase will social network research conducted by studying actors linked together by social relations. This will be achieved through net mapping exercise to understand, discuss, and visualize how various actors influence pneumonia related outcomes through technical and financial links. Data will be analyzed through the Organizational Risk Analyzer (ORA) which is a meta-network assessment and analysis tool. This study will be the first of its kind for under-five pneumonia and will guide policy makers for creating effective solutions to combat the disease.

DETAILED DESCRIPTION:
Despite the availability of standard pneumonia management guidelines and multiple global efforts, pneumonia continues to be the leading killer of children under five, accounting to around 17% of the total under five deaths globally. It has been estimated that annually there are around 120 million episodes of pneumonia among children with around 14 million progressing to severe episodes. Out of these cases, close to 1.3 million children die with 81% of these deaths occurring under 2 years of age. 52% of these deaths occur in the Sub-Saharan region and South Asia with main contributions from India, Nigeria, Congo, Pakistan and Afghanistan. In Pakistan, pneumonia contributes to 16% of under-five mortality in the country with annually around 65,000 children dying due to this disease; a status unchanged for more than a decade.

In order to reduce pneumonia related morbidity and mortality, World Health Organization (WHO) and United Nations International Children's Emergency Fund (UNICEF) have developed multiple action/ intervention plans. This includes initiatives like the Integrated Global Action Plan for the Prevention and Control of Pneumonia and Diarrhea, Global Strategy for Women's and Children's Health, Committing to Child Survival, Global Vaccine Action Plan etc. All these initiatives/interventions focus on a unified goal of "ending preventable deaths". They bring together critical interventions to promote practices to save lives of children, to create healthy environments and to have access to appropriate preventive and treatment measures. Pakistan, among other countries, has been actively involved in various related forums on prevention and management of pneumonia. But for best outcomes at national level, such initiatives need to be supported by appropriate policies/strategies because policies entail political and strategic support for best management and care. Also needed is engagement by regional governance structures, including roles such as coordination, funding, and guidelines for policy development.

Pakistan has launched multiple national programs in line with these global initiatives at various periods of time. These programs include the National Acute Respiratory Illness (ARI) control program which was launched in 1989 with the main objectives of reducing severity and mortality due to pneumonia and rationalize the use of antimicrobial and other drugs for treatment of ARI. WHO soon realized that this disease centric narrow approach has not been able to achieve its desired objectives. Therefore, it developed a more integrated approach and launched it globally as Integrated Management of Childhood Illnesses (IMCI) launched in Pakistan in 1998. The approach in IMCI focused on improving case management skills of health workers, strengthening the health system, and addressing family and community practices. Duplicity was very much evident from the fact that ARI existed as an independent program and was also part of the IMCI package. Between 2004-2010 The Pakistan Initiative for Mothers and Newborns (PAIMAN), a United States Agency for International Development (USAID) funded project was undertaken which focused on improving the status of maternal and newborn health in 24 districts across the four provinces and Azad Jammu and Kashmir (AJK) in Pakistan. ARI was an important component in that project. Thereafter, a national Maternal, Neonatal and Child Health program (MNCH) was launched in 2010 funded mainly by Department for International Development (DFID) focused on strengthening of management and organization mechanism of healthcare delivery systems which ended after 5 years.

This shows that there has been a constant flow of ARI related program initiation and termination which could be attributed to the unsteady health policy environment of Pakistan markedly influenced by the unsteady political environment. Before 2011, the health ministry at the federal level was responsible for policy development, implementation, monitoring and surveillance. In June 2011 in wake of the 18th amendment of the national constitution, this National Health Ministry was devolved. This led to the shift of certain responsibilities from the federal level to the provinces. As a result, health policy formulation, planning along with service delivery was devolved to the provinces leading to differences in health outcomes across the country. Considering the development of all these programs/strategies/policies has been influenced by various stakeholders including the ministry, academicians, researchers, physicians, and development partners, it is, therefore, important to understand how different actors come together and influence policy making and implementation. This could assist in exploring the existing policy support for reducing pneumonia related morbidity and mortality and thus underpin recommendations for improving the status.

Primary Objective

* To identify and analyse pneumonia related policies/ strategies in Pakistan for children under five.
* To identify key stakeholders who shape under five pneumonia related policy environment, through technical and/or financial contributions.

Secondary Objectives

* To identify how under five pneumonia related policies are developed and implemented in Pakistan.
* To identify barriers and/or facilitators for under five pneumonia related policy development and implementation

Methodology:

A descriptive study design will be used for this study which will be conducted through pneumonia related policy "content analysis" along with net map activities and in depth interviews to collect both qualitative and quantitative data on the stakeholders involved and their level of support and influence to the cause (stakeholder analysis). The basic purpose of coupling policy content analysis with stakeholder analysis is to correlate ground realities with what has been mentioned in the policies/strategies.

Content Analysis:

We will use Walt and Gilson's framework for policy analysis, which focuses on policy content, actors, context, and process (agenda-setting, policy development, implementation) as indicated in Figure 1[17-19]. Walt and Gilson developed a policy analysis framework specifically for health, although its relevance extends beyond this sector. They noted that health policy research focused largely on the content of policy, neglecting actors, context and processes. Their policy triangle framework considers how all four of these elements interact to shape policy-making. The framework has influenced health policy research in a diverse array of countries, and has been used to analyse a large number of health issues, including mental health, health sector reform, tuberculosis, reproductive health and antenatal syphilis control.The aim of this component is to map the pneumonia related policies and strategies in Pakistan. We will first develop a matrix to guide the data collection process. This matrix will be developed through a mind mapping exercise to identify relevant policy document types. These document types could be:

* Government strategic plans (5-10 year)
* Health ministry action plan
* Any legislation
* Any national or provincial pneumonia related strategies/guidelines
* General program guidelines with pneumonia as a component
* Any training guidelines on pneumonia
* Any facility guidelines
* Any community intervention guidelines
* Any monitoring guidelines

Relevant documents will then obtained. We plan to source documents from government websites, government archives, and through requests to Ministry of Health officials (and those from related Ministries), development partners, and researchers involved in pneumonia related research in the past. We will acquire policies from the provinces of Punjab, Sindh, Baluchistan and Khyber Pakhtukhuwa (KPK). All the relevant documents will then be explored for the information as indicated in the matrix. For each policy document, we will note:

1. Any mention of pneumonia (as per matrix)
2. Name of Policy
3. Year of release
4. Released by (e.g. which ministry)
5. Component/section of the document with relevant information

All documents will be copied and retained.

Stakeholder Analysis:

Qualitative Interviews:

In this phase of research, we will identify how pneumonia related policies are conceptualized, developed, implemented and delivered through a qualitative approach. This will be accomplished through "grounded theory" by conducting in depth interviews from key informants. This will be explored through policy makers, program managers, academicians, researchers and healthcare providers. This means that we will draw on both 'top-down' and 'bottom-up' theories of implementation incorporating the perspectives of both health policy makers and implementer of the policy. The policy content analysis will also guide the development of the interview guides. The content of the interviews will be (not limited to):

* A brief on the roles and responsibilities of the respondents
* Their knowledge of pneumonia related policy environment
* How such policies/strategies have been/are developed
* What has the respondents' role been in the development and implementation of such policies
* What are barriers and facilitators of policy development and implementation
* Who are the key stakeholders involved in influencing pneumonia related policies
* What are the key recommendations for sustainable implementation of these policies to reduce pneumonia related morbidity and mortality in the long run.

Respondents will be those spread across the country and focus will be in post devolution era. But if highly valuable information is being provided by respondents on the pre devolution era then that will also be noted. This will help in assessing difference among provinces as well.

Net Mapping Activities:

We will use the Net-Map method developed by International Food Policy and Research Institute (IFPRI) to map and analyze information regarding stakeholder influence. Net mapping is a part of social network research. We shall be using this technique also based on prior experience in health policy research. A social network is a group of actors that are linked together by a set of social relations. These relations describe the ties of a specific kind among the actors of the network. The key principles within social research are:

(i) actors and their actions in a social network viewed as interdependent rather than independent, autonomous units; and (ii) relational ties between actors as channels for transfer of resources (either material or non-material. The location of an actor inside a social network can be an indicator of the strength of ties associated with that actor. Moreover, net mapping provides both a visual and a mathematical analysis of network relations among actors within that network.

These activities will be group based interviews whereby upon identification of key stakeholder/ groups through the qualitative approach, relevant stakeholders will be recruited upon taking consent and these group activities will be conducted in each province. A net map interview guide will be developed focusing on the following research questions:

* Who are the influential stakeholders who provide technical contributions in pneumonia related policy environment in Pakistan.
* Who are the influential stakeholders who provide financial contributions in pneumonia related policy environment in Pakistan.
* What is their level of influence in pneumonia related policy environment in Pakistan where influence is referred to as formal supervision, funding, technical information, advice, advocacy and pressure, but might go beyond the links mentioned above, e.g. Influence because one is respected.
* What is their level of support in pneumonia related policy environment in Pakistan.

Each group activity will start by listing down the names of relevant stakeholders, referred to as actors, who provide technical and/or financial support for pneumonia related policy environment in Pakistan. For drawing maps, we will first consider Technical support which is defined as formal exchange of technical support (training, technical guides, equipment, staff/consultant (pres elected), information, research evidence, routine data, and field experience/case studies). This will be followed by Funding support which is defined as exchange of funds or in-kind support (this could be funding or supplies for programs or staff employed by the recipient, or budget provision). For both kind of supports we will ask first about the technical support that the actor receives, then who the actor provides it to ("from whom?", then "to whom?"). Arrows will be drawn between actors and their support links whereby a different color will be used for technical and financial links. After drawing the links, level of influence will be identified against each actor which could be high or low indicated as positive or negative. This will be followed by identifying the level of support which every actor has on the cause. The rate used is supportive, not supportive and neutral.

Descriptive Analysis Approach. The steps involved in synthesis will include development of a theoretical model revolving around pneumonia related policy environment, preliminary synthesis using the matrix, and exploring associations in the data. This approach will enable us to consider specific policy content within the broader policy context.

Data Analysis:

In depth interviews will be analysed through development of themes and sub themes which will be drawn from the framework used in content analysis with particular emphasis on the type of actors and their role in the process, the structure and content of the policies and experiences of implementation and suggestions of those in the system. Qualitative and quantitative data of the net map activities will be triangulated. The quantitative data will be analysed using ORA (Organizational Risk Analyzer), specialized software meant for analysis of net map data.

ELIGIBILITY:
Inclusion Criteria:

* Those respondents who are directly involved or knowledgeable about pneumonia related policy environment in the country/province.
* Respondents who consent to participate in the study.
* Respondents belonging to Sindh, Punjab, Baluchistan, KPK and Islamabad.

Exclusion Criteria:

* Respondents belonging to Gilgit-Baltistan (GB), Azad Jammu and Kashmir (AJK) and Federally Administered Tribal Area (FATA). Reasons of their exclusion are newly developed governance system (GB), separate governance (AJK) and security threat (FATA).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For the qualitative phase of interviews and focus group discussions, purposeful sampling will be employed and the sample size will be based on the point of theoretical saturation, although at least 20 interviews will be conducted (4 in each of the five administrative divisions; Punjab, Sindh, Baluchistan, KPK and Federal capital). The type of respondents for the in depth interviews would be policy makers, program managers, project coordinators (national or provincial), academicians, researchers, practitioners etc.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Identification of Pneumonia Policy Formation in Pakistan | 12 months
  To identify and analyse pneumonia related policies/strategies in Pakistan for children under five. A matrix would be developed to assess all relevant national and governmental policies related to pediatric pneumonia in Pakistan. Descriptive content analysis would be conducted for national policies on acute respiratory illness (both federal and provincial).
Facilitators and barriers for under five pneumonia related policy development and implementation | 6 months
  In depth interviews of key stakeholders will be conducted to assess the facilitators and barriers to under five pneumonia related policy development and implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tabish Hazir, MBBS, FRCPCH, Principal Investigator — Maternal, Neonatal and Child Health Research Network
Locations (1):
- Maternal, Neonatal and Child Health Research Netork, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided